CLINICAL TRIAL: NCT06224426
Title: Oxygenation Targets for Endovascular Therapy in Acute Ischemic Stroke Patients (Oxy-TARGET)
Brief Title: Oxygen Concentration Target in Stroke Endovascular Treatment
Acronym: Oxy-TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Lead Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zkd20231121
Record Dates: First submitted 2023-12-17; First posted 2024-01-25 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke
Keywords: Endovascular therapy; Acute ischemic stroke; Normobaric hyperoxia; Early neurological improvement; General anesthesia
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normobaric high-concentration oxygen (NBHO) group (Experimental): After preoxygenating (FiO2=100%, 6 L/min) with a face mask for 3 min, patients will be sequentially administered intravenous sufentanil 0.2 µg/kg followed by propofol 2 mg/kg. Once the eyelash reflex was absent, all patients received 0.6 mg/kg rocuronium, with an endotracheal tube inserted approximately 90 seconds later. Mechanical ventilation is set to volume-controlled ventilation (VCV) mode, fresh gas flow 4 L/min, tidal volume (Vt) 6-8 ml/kg, respiratory rate (RR) 12-14 breaths/min, and positive end-expiratory pressure (PEEP) 5 cmH2O. End-tidal carbon dioxide (PetCO2) will be continuously monitored, maintaining it between 35-40 mmHg. Based on group allocation, the NBHO group will adjust the FiO2 at 80% throughout the surgery. Anesthesia will be maintained through total intravenous anesthesia, continuously infusing remifentanil 0.05-0.1 µg/kg/min and propofol 4-6 mg/kg/min, with intermittent 10 mg rocuronium as needed.
  Interventions: Other: Normobaric high-concentration oxygen
- Normobaric low-concentration oxygen (NBLO) group (Experimental): After preoxygenating (FiO2=100%, 6 L/min) with a face mask for 3 min, patients will be sequentially administered intravenous sufentanil 0.2 µg/kg followed by propofol 2 mg/kg. Once the eyelash reflex was absent, all patients received 0.6 mg/kg rocuronium, with an endotracheal tube inserted approximately 90 seconds later. Mechanical ventilation is set to volume-controlled ventilation (VCV) mode, fresh gas flow 4 L/min, tidal volume (Vt) 6-8 ml/kg, respiratory rate (RR) 12-14 breaths/min, and positive end-expiratory pressure (PEEP) 5 cmH2O. End-tidal carbon dioxide (PetCO2) will be continuously monitored, maintaining it between 35-40 mmHg. Based on group allocation, the NBLO group will adjust the FiO2 at 30% throughout the surgery. Anesthesia will be maintained through total intravenous anesthesia, continuously infusing remifentanil 0.05-0.1 µg/kg/min and propofol 4-6 mg/kg/min, with intermittent 10 mg rocuronium as needed.
  Interventions: Other: Normobaric low-concentration oxygen

INTERVENTIONS:
Other: Normobaric high-concentration oxygen — During endovascular therapy, eligible participants will receive FiO2=80% through endotracheal intubation, with a gas flow rate set at 4 L/min.
  Arms: Normobaric high-concentration oxygen (NBHO) group
Other: Normobaric low-concentration oxygen — During endovascular therapy, eligible participants will receive FiO2=30% through endotracheal intubation, with a gas flow rate set at 4 L/min.
  Arms: Normobaric low-concentration oxygen (NBLO) group

SUMMARY:
The goal of this clinical trial is to compare the effects of different concentrations of normobaric oxygen on early neurological improvement in acute ischemic stroke (AIS) patients receiving endovascular therapy (EVT). The main questions it aims to answer are:

* Evaluating the impact of normobaric high-concentration oxygen versus low-concentration oxygen on early neurological function after EVT.
* Evaluating the safety of high and low normobaric oxygen concentration in patients with ischemic stroke.

Participants will (1) receive EVT under general anesthesia; (2) be randomly assigned 1:1 to receive oxygen therapy with FiO2=80% or FiO2=30% through endotracheal intubation during the operation, and the gas flow rate was set at 4L /min.

DETAILED DESCRIPTION:
The optimal fraction of inspired oxygen (FiO2) during EVT under general anesthesia is currently uncertain. This is a randomized controlled trial (RCT) designed to assess the impact of normobaric high-concentration oxygen versus low-concentration oxygen on early neurological function following EVT. It is a prospective, open-label, parallel-design RCT planned to be conducted at Beijing Tiantan Hospital, Capital Medical University. It is anticipated that 200 cases of AIS patients undergoing EVT under general anesthesia will be consecutively enrolled from 2024 to 2026. Eligible participants will be randomly assigned in a 1:1 ratio. After general anesthesia induction, patients will receive continuous inhalation of oxygen with either FiO2=80% or FiO2=30% through endotracheal intubation until the end of the procedure, with a gas flow rate set at 4 L/min. The positive end-expiratory pressure (PEEP) is uniformly set to 5 cmH2O to balance its effect on pulmonary oxygen delivery. The primary outcome will be the occurrence of early neurological improvement (NIHSS score of 10 points 24±2 hours after EVT). Safety outcomes include potential adverse events such as site infection, three-month mortality, etc.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years.
2. Anterior circulation occlusive stroke is confirmed by CT angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography (DSA), and occlusions of intracranial internal carotid artery (ICA) or M1 segment of the middle cerebral artery (MCA) were involved.
3. NIHSS score at admission: 6-20.
4. Randomization can be completed within 24 hours after stroke onset.

Exclusion criteria

1. Stroke onset within 6-24 hours with a CT perfusion imaging (CTP)-assessed mismatched area<15 ml.
2. Presence of anemia, defined as hemoglobin levels o below 120 g/L in men and below 110 g/L in women.
3. Pre-stroke modified Rankin scale (mRS) score ≥2.
4. Complicated by severe agitation and seizures.
5. Evidence of intracranial hemorrhage at admission.
6. Presence of chronic obstructive pulmonary disease, asthma, or other respiratory conditions, or requirement for daily supplemental oxygen or mechanical ventilation.
7. Baseline arterial blood gas analysis indicating impaired gas exchange: PaO2 < 60 mmHg on room air, or oxygenation index (PaO2/FiO2) < 300 mmHg with supplemental oxygen.
8. Emergency chest CT reveals significant pulmonary parenchymal infection.
9. An oxygen mask or ventilator must be used before anesthesia to maintain a SpO2≥94%.
10. Loss of airway protective reflex or vomiting aspiration upon admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of early neurological improvement (ENI) | 24±2 hours after EVT
  ENI is defined as an NIHSS score of <10 points at 24±2 hours after EVT

SECONDARY OUTCOMES:
ΔNIHSS at 24±2 hours after EVT | 24±2 hours after EVT
  baseline NIHSS score - NIHSS score at 24±2 h
the final infarct volume | 72 hours post-randomization
  After collecting cranial CT images, the infarct volume was delineated using ITK-SNAP software.
early neurological deterioration (END) | 1 day after reperfusion therapy
  an increase of ≥4 from the baseline NIHSS score on day 1 after reperfusion therapy in AIS patients
Postoperative pulmonary complications | within 7 days after endovascular therapy
  defined as a composite measure encompassing pulmonary infections, atelectasis, pleural effusion, respiratory failure, bronchospasm, and pneumothorax
overall mRS distribution at 90 days | 90 days after stroke onset
  modified Rankin scale (mRS) scores are distributed between 0 and 6
favorable functional outcome | 90 days after stroke onset
  an mRS score of 0-2 at 90 days

OTHER OUTCOMES:
Postoperative baseline PaO2 | From the end of the intervention procedure until the time just before the tracheal tube is removed.
  Arterial partial oxygen pressure based on arterial blood gas
Postoperative baseline oxygenation index | From the end of the intervention procedure until the time just before the tracheal tube is removed.
  oxygenation index=PaCO2/FiO2
symptomatic ICH | 24±12 hours after EVT
  defined as the presence of hemorrhage on CT at 24±12 h accompanied by an NIHSS score increase≥4
all-cause mortality at 90 days | 90 days after stroke onset
  deaths from any cause during the 3-month follow-up period
stroke-related death | within 7 days after endovascular therapy
  typically defined as death directly attributable to the stroke and its complications, encompassing but not limited to severe cerebral edema, brain herniation, infections, cardiac diseases, pulmonary embolism, and deep vein thrombosis occurring during the acute phase of AIS

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, Ph.D, Study Director — Department of Anesthesiology, Beijing TianTan Hospital, Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Z, Zhang K, Wu Y, Wang X, Zhang Z, Hou X, Jian M, Wang Y, Liu H, Wang A, Han R, Liang F. Oxygenation targets for endovascular therapy in acute ischemic stroke patients (Oxy-TARGET): protocol for a single-centre, open-label randomised controlled trial. BMJ Open. 2025 Jan 4;15(1):e086234. doi: 10.1136/bmjopen-2024-086234. PMID 39755573